CLINICAL TRIAL: NCT06042699
Title: Kids With Iron Deficiency and Scoliosis (KIDS) Study
Brief Title: Kids With Iron Deficiency and Scoliosis
Acronym: KIDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Lisa Eisler, Assistant Professor of Anesthesiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AAAU2577; K23GM152933-01 (NIH)
Record Dates: First submitted 2023-09-12; First posted 2023-09-18 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Adolescent Idiopathic Scoliosis; Neuromuscular Scoliosis; Perioperative/Postoperative Complications; Iron Deficiencies; Anemia; Spinal Fusion; Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Postoperative Complications; Iron Deficiencies; Anemia; Postoperative Cognitive Complications | interventions — ferrous sulfate

STUDY DESIGN:
Intervention Model Description: Double blind placebo-controlled randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo tablets will be indistinguishable from iron tablets. Group allocation will not be accessible to participants, care providers, investigators, or outcomes assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Oral ferrous sulfate (Experimental): Participants will receive oral ferrous sulfate tablets, 325mg (65mg elemental iron). Tablets are to be taken once daily for 3-6 months prior to surgery as time allows.
  Interventions: Dietary Supplement: Oral ferrous sulfate
- Oral placebo tablets (Placebo Comparator): Participants will receive placebo tablets. Tablets are to be taken once daily for 3-6 months prior to surgery as time allows.
  Interventions: Dietary Supplement: Oral placebo tablet
- Observational follow-up (No Intervention): Participants who do not qualify for randomization may be invited to complete study measures through postoperative follow-up as part of an observational study.

INTERVENTIONS:
Dietary Supplement: Oral ferrous sulfate — Oral ferrous sulfate 325mg is used as a dietary supplement providing 65mg elemental iron.
  Arms: Oral ferrous sulfate
Dietary Supplement: Oral placebo tablet — Oral placebo tablet provided as placebo comparator.
  Arms: Oral placebo tablets

SUMMARY:
This study is a randomized controlled trial of preoperative oral iron supplementation, to identify whether iron deficiency is a modifiable risk factor for adverse surgical outcomes such as red blood cell transfusion and diminished postoperative cognitive and physical capacity in adolescents undergoing scoliosis surgery.

Research Question(s)/Hypothesis(es):

Primary

* Iron supplementation will reduce the incidence of perioperative RBC transfusion in iron deficient scoliosis patients undergoing spinal fusion.

Secondary

* Iron supplementation will reduce postoperative neurocognitive functional declines in iron deficient scoliosis patients undergoing spinal fusion.
* Iron supplementation will improve patient-reported physical functioning in iron deficient scoliosis patients undergoing spinal fusion.

DETAILED DESCRIPTION:
Adolescents undergoing spinal fusion surgery for scoliosis are poised to benefit from preoperative iron supplementation. Spinal fusion carries a risk of large surgical blood losses and perioperative red blood cell transfusion, which are associated with adverse outcomes in this population. These patients are mostly adolescent females, a group more susceptible to iron deficiency and resulting anemia at baseline due to iron losses with menses, and who suffer an additional insult to iron stores during surgery. Nevertheless, iron status is not routinely monitored in this setting and there is no standard of care for preoperative iron supplementation. Iron is a nutritionally essential trace element important not only for red blood cell production, but also for muscle function and neurotransmitter synthesis and signaling. Therefore, the treatment of preoperative iron deficiency is an important target for optimizing hemoglobin prior to surgery, reducing transfusion rates and associated complications such as alloimmunization, and improving patient outcomes. On its own and as the primary cause of anemia, iron deficiency was identified by the investigator's team as the only risk factor for transfusion which is modifiable preoperatively.

In addition, iron supplementation is shown to alleviate impairments of physical and cognitive capacity associated with even mild forms of iron deficiency in adolescent females. A pilot study conducted at the investigator's institution identified iron deficiency in 36% of scoliosis patients prior to surgery, with preoperative iron status highly correlated with iron status during surgical recovery. Consequently, the investigator plans to examine iron deficiency as a modifiable risk factor for transfusion and impaired postoperative cognitive and physical capacity in this vulnerable population. Previous trials of brief iron interventions in high-risk adult surgical patients, mostly with unknown iron status, do not inform the care of iron deficient adolescents and were not designed to address postoperative functional outcomes. This study will therefore perform a single-center randomized controlled trial in which adolescents with scoliosis will be screened for iron deficiency (n = ~275), and iron-deficient adolescents with scoliosis (n = ~90) will be randomized to a preoperative regimen of daily oral iron or placebo, to test the hypotheses that preoperative iron supplementation 1) reduces the rate of red blood cell transfusion, 2) improves postoperative neurocognition compared to a preoperative baseline, and 3) improves patient-reported physical functioning during recovery. Results will ultimately improve outcomes in this vulnerable pediatric population and provide evidence for patient blood management approaches to reduce transfusions amid recent severe blood shortages.

ELIGIBILITY:
Inclusion Criteria:

1. 10-26 years old;
2. diagnosis of scoliosis or kyphosis;
3. self-reported ability to swallow a tablet;
4. spinal fusion procedure planned approximately 6 to 24 weeks from an orthopedic surgical clinic visit at which patient agrees to phlebotomy for screening blood work;
5. serum ferritin less than or equal to 25 µg/L.

Exclusion Criteria:

1. taking or planning to take iron-containing supplement on patient's own volition, and not willing to stop for duration of study;
2. taking or planning to take iron-containing supplement as prescribed or recommended under the care of a physician;
3. Hg <10mg/dL if post-menarchal, Hg < 11 if premenarchal or male
4. C-reactive protein > 10 mg/L
5. receiving nutritional support by report in the medical chart;
6. self-reported history of hypersensitivity reaction to iron-containing supplements;
7. self-reported history of or suspected non-iron deficient hematologic disorder;
8. self-reported history of iron overloaded state such as hereditary hemochromatosis or hemosiderosis;
9. objection to receiving red blood cell transfusions;
10. current pregnancy (by self-report);
11. prisoners;
12. patient or parent decides against study participation.

Ages: 10 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 275 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of perioperative RBC transfusion in iron deficient scoliosis patients undergoing spinal fusion | 4 to 30 days
  The patients that received a red blood cell transfusion either during procedure or postoperatively during t surgical hospitalization will be tallied.

SECONDARY OUTCOMES:
Percentage of Patients that experienced postoperative decline in neurocognitive function | 3-6 months
  The Cognitive Battery of the NIH Toolbox is a brief, valid, and reliable instrument designed to provide outcome measures in epidemiologic and longitudinal research that can be used for comparisons across a wide range of studies and populations. Individual measure scores in the battery reflect Executive Function, Attention, Verbal and Nonverbal Memory, Language, Processing Speed, and Working Memory, yielding composite score. A decline of function is measured by comparing the mean change from baseline in the Cognitive Function Composite Scores in the study groups. Higher raw scores reflect higher function in the tested domains, and age-adjustment is then performed such that Age-Corrected Standard scores compare the score of the test-taker to those in the NIH Toolbox nationally representative normative sample at the same age, where a score of 100 indicates performance that was at the national average for the test-taking participant's age.
Percentage of patients that experienced postoperative decline in self-reported physical capacity | 3-6 months
  The PROMIS pediatric measures are a NIH Roadmap initiative to provide access to valid and reliable self-reported measures of health-related quality of life in children and adolescents. The PROMIS measures are scored on a T-score metric with a mean of 50 and SD of 10 in the general population in the United States. Higher PROMIS symptom scores indicate increased symptom burden, and higher PROMIS function scores indicate increased functioning. Decline would be identified through a mean change (decrease) from baseline in the Physical Functioning - Mobility scores; with secondary hypotheses for Physical Functioning - Upper Extremity, Physical Activity, and Fatigue.
Volume of perioperative RBC transfusion | 4 to 30 days
  The volume that each patient receives either during procedure or postoperatively during surgical hospitalization will be summed and average calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa D Eisler, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared.